CLINICAL TRIAL: NCT02120209
Title: Nurse Screening Tool for Fall Risk : Prediction of Falls in Older Inpatients Hospitalized at Angers University Hospital
Brief Title: Prediction of Falls in Older Inpatients Hospitalized at Angers University Hospital
Acronym: EPRIC
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2013/24
Record Dates: First submitted 2014-04-17; First posted 2014-04-22 (Estimated); Last update posted 2014-04-22 (Estimated); Status verified 2014-04

CONDITIONS: to Elaborate a New Simple Clinical Tool for the Risk of Falls Among Older Inpatients.
Keywords: assessment; falls; older adults; prediction scale; standardized declaration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of this study is to elaborate a new simple clinical tool for the risk of falls among older inpatients.

DETAILED DESCRIPTION:
Falling is a common event within hospitals, with a rate calculated between 2.9-13 per 1,000 bed-days . Falls lead to prolonged length of hospital stays (LHS). The first step of an efficient and cost-effectiveness strategy of fall prevention is the screening of individuals at higher risk of falls. Recently, a brief geriatric assessment (BGA) composed of a few number of items has demonstrated to successfully predict the risk of prolonged LHS (5). We hypothesized that the use of the BGA items would make it possible to predict the occurrence of falls among older inpatients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* participants who did not issue opposition to participation in the study
* Patients hospitalized at the University Hospital of Angers in acute care units participating in study
* Being affiliated to a social security regime

Exclusion Criteria:

* Opposition to the use of information collected for research purposes.
* Age < 65 years

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients hospitalized in acute care units participating in study in Angers University Hospital with respect to the eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Actual)
Dates: Start 2013-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Clinical characteristics (i.e., Brief geriatric assessment items) | recorded at baseline when older adult were admited to acute care units.

SECONDARY OUTCOMES:
Occurrence of falls | assessed between 2 and 21 hospitalization days
Number of falls | assessed between 2 and 21 hospitalization days
Severity of falls | assessed between 2 and 21 hospitalization days

CONTACTS AND LOCATIONS:
Locations (1):
- University Memory Center, Angers University Hospital, Angers, Pays de la Loire Region, France